CLINICAL TRIAL: NCT02250443
Title: An Open-label, Long-term Study to Evaluate the Safety and Tolerability of BYM338 in Patients With Sporadic Inclusion Body Myositis
Brief Title: Study of Long-term Safety, Efficacy Tolerability of BYM338 in Patients With Sporadic Inclusion Body Myositis
Acronym: BYM338
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBYM338X2205E1
Record Dates: First submitted 2014-03-20; First posted 2014-09-26 (Estimated); Results first posted 2018-04-10 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2019-03

CONDITIONS: Sporadic Inclusion Body Myositis (sIBM)
Keywords: Inclusion Body Myositis (IBM)
MeSH Terms: conditions — Myositis, Inclusion Body | interventions — bimagrumab

ARMS (1):
- BYM338 (Experimental): BYM338 Group
  Interventions: Drug: BYM338 (Bimagrumab)

INTERVENTIONS:
Drug: BYM338 (Bimagrumab)

SUMMARY:
This study is an open-label, long-term study for those patients who participated in the prior proof-of-concept protocol, in which the preliminary efficacy for BYM338 in patients with sIBM was demonstrated after a single 30 mg/kg i.v. dose of BYM338. This study is designed to confirm the efficacy, safety and tolerability of BYM338 in sIBM with long-term dosing. However due to lack of efficacy in patients with sIBM, the study was terminated early.

DETAILED DESCRIPTION:
This is a non-confirmatory, multicenter, open-label, non-randomized trial which will extend active treatment to those patients that participated in the preceding proof-of-concept study (CBYM338X2205) in order to collect long-term safety and tolerability data. Up to 14 patients with sIBM will be invited to enroll into the study to receive BYM338 open-label for a period of approximately 3 years or until BYM338 is commercially available, whichever comes first. The study consists of a maximum 28-day screening period, a 5-day baseline period, and a treatment period consisting of the site visits at 4-week intervals for treatment administration, safety and pharmacokinetic follow-up. All patients will be administered a medium level i.v. BYM338 dose regardless of their treatment allocation in the prior study.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained before any assessment is performed.
* Patients who participated in the CBYM338X2205 study. A patient is defined as participating in the study if they were enrolled and received study medication.
* Able to communicate well with the investigator, to understand and comply with the requirements of the study.

Exclusion Criteria:

* Patients for whom the treating physician considers it inappropriate for continuation into the study, including consideration of physical and laboratory assessment of the patient at screening.
* Patients who were non-compliant or demonstrated a serious protocol deviation in the previous study.
* Use of other investigational drugs at the time of enrollment, within 30 days or 5 half-lives of enrollment, or until the expected PD effect has returned to baseline, whichever is longer; or longer if required by local regulations.
* History of hypersensitivity to any of the study drugs or to drugs of similar chemical classes
* Swallowing difficulty or other reason that precludes adequate intake of energy and protein, defined as at least 20 kcal/kg/day and 0.6 g protein/kg/day as determined by the investigators assessment.
* On the Columbia-Suicide Severity Rating Scale, a score of 4 or 5 on the Suicidal Ideation item or any "yes" on the Suicidal Behavior item that is related to suicidal behavior occurring during the last 2 years.
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test.
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, must use highly effective contraception during the study and for 5 half-lives (14 weeks) after stopping treatment. Highly effective contraception is defined as either:

  1. Total abstinence: When this is in line with the preferred and usual lifestyle of the subject. [Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception].
  2. Sterilization: have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.
  3. Male partner sterilization (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate). [For female study subjects, the vasectomized male partner should be the sole partner for that patient].
  4. Use of a combination of any two of the following (a+b or a+c or b+c):

  <!-- -->

  1. Use of oral, injected or implanted hormonal methods of contraception.
  2. Placement of an intrauterine device (IUD) or intrauterine system (IUS).
  3. Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository.

In case of use of oral contraception women should have been stable on the same pill for a minimum of 3 months before taking study treatment. Postmenopausal females must have had no regular menstrual bleeding for at least one (1) year prior to initial dosing. Menopause will be confirmed by a plasma FSH level of > 40 IU/L (or as determined by the cut off used by the local clinical laboratory) at screening. Female patients who report surgical sterilization must have had the procedure at least six (6) months prior to initial dosing. Surgical sterilization procedures should be supported with clinical documentation made available to the sponsor and noted in the Relevant Medical History / Current Medical Conditions section of the eCRF. All female patients must have negative pregnancy test results at screening and baseline.

* Use of oral beta agonists, oral corticosteroids, androgens or androgen inhibitors (including LHRH agonists), or intravenous gamma globulin (IVIG) within the previous 6 months. Short-term corticosteroids for unrelated indications, defined as < 20 mg/d for < 30 days and ending at least 60 days prior to screening, are acceptable.
* Patients with known bleeding disorders, or who are under treatment with anti-coagulants.
* A presence or history of clinically relevant ECG abnormalities, or including but not limited to Long QT syndrome, ischemic changes that cannot be shown to be stable for at least 6 months by previous ECG, or 2nd degree Mobitz II or 3rd degree heart block.
* History of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases.
* Significant illness which has not resolved within two (2) weeks prior to initial dosing.
* A positive HIV, Hepatitis B surface antigen or Hepatitis C test result. No additional exclusions may be applied by the investigator, in order to ensure that the study population will be representative of all eligible patients.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-03-11 (Actual); Primary Completion 2016-08-23 (Actual); Study Completion 2016-08-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- United States (2):
  - Novartis Investigative Site, Phoenix, Arizona
  - Novartis Investigative Site, Boston, Massachusetts

REFERENCES:
- [Derived] Sivakumar K, Cochrane TI, Sloth B, Ashar H, Laurent D, Tanko LB, Amato AA. Long-term safety and tolerability of bimagrumab (BYM338) in sporadic inclusion body myositis. Neurology. 2020 Oct 6;95(14):e1971-e1978. doi: 10.1212/WNL.0000000000010417. Epub 2020 Jul 20. PMID 32690797
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=184

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Due to lack of efficacy in patients with sIBM, the study was terminated early.
Period: Overall Study
Arm/Group | BYM338
Started | 10
Completed | 0
Not Completed | 10
Not completed — Administrative problems | 7
Not completed — Adverse Event | 3

BASELINE CHARACTERISTICS:
Arm/Group | BYM338
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.1 (10.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability
Description: Any Adverse Event was defined as occurrence of any symptom regardless of intensity grade, Serious Adverse Event (SAEs) assessed as medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in persistent or significant disability/incapacity
Time Frame: Up to 29 month
Population: safety analysis set - included all patients that received at least one dose of study drug. No statistical analysis provided for Number of Participants Who Experienced Adverse Events (AEs) and Serious Adverse Events (SAEs) During this extension study
Measure: Number; unit: Participants
Arm/Group | BYM338
Number analyzed (Participants) | 10
Participants
  Death | 0
  Serious adverse events (SAE) | 2
  Adverse Events (AE) | 10

2. Secondary Outcome: Changes From Baseline in Lean Body Mass (LBM) by Dual-Energy X-ray Absorptiometery (DXA)
Description: To assess the effect of multiple doses of BYM338 on lean body mass as measured by DXA in terms of change from baseline.
Time Frame: Baseline, Day 1, 57, 113, 169, 365, 533, and day 729
Population: Pharmacodynamics (PD) analysis set: Patients with evaluable PD parameter data
Measure: Mean (Standard Deviation); unit: Percentage Change in LBM
Arm/Group | BYM338
Number analyzed (Participants) | 10
Percentage Change in LBM
  Day 1 | 0 (0)
  Day 57 | 4.292 (2.7480)
  Day 113 | 5.552 (3.6066)
  Day 169 | 7.463 (4.5687)
  Day 365 | 6.919 (2.9669)
  Day 533: number analyzed (Participants) | 8
  Day 533 | 6.885 (3.7894)
  Day 729: number analyzed (Participants) | 1
  Day 729 | 0.727 (NA) — NA- Not available, standard deviation is not evaluable when n=1

3. Secondary Outcome: Pharmacokinetics (PK) Parameter of Cmin From Multiple i.v. Dosing
Description: To obtain pharmacokinetic data from multiple i.v. dosing of BYM338 in this patient population. Pre-dose, 30 mins & 4 hours post-dose on Day 1. Pre-dose only on each subsequent administration
Time Frame: Day 29, 85, 169, 253, 337, 421, 505, 589, 673, 757, 1177
Population: Pharmacokinetics (PK) Analysis set: Patients with available PK data and no protocol deviations with relevant impact on PK data
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | BYM338
Number analyzed (Participants) | 10
ng/mL
  Day 29 (n=10) | 13.4 (5.01)
  Day 85 (n=10) | 24.1 (13.1)
  Day 169 (n=10) | 26.3 (15.9)
  Day 253 (n=9): number analyzed (Participants) | 9
  Day 253 (n=9) | 28.8 (12.1)
  Day 337 (n=10) | 24.4 (14.6)
  Day 421 (n=9): number analyzed (Participants) | 9
  Day 421 (n=9) | 24.5 (11.5)
  Day 505 (n=8): number analyzed (Participants) | 8
  Day 505 (n=8) | 28.3 (10.6)
  Day 589 (n=6): number analyzed (Participants) | 6
  Day 589 (n=6) | 39.8 (30.2)
  Day 673 (n=2): number analyzed (Participants) | 2
  Day 673 (n=2) | 20.5 (1.98)
  Day 757 (n=1): number analyzed (Participants) | 1
  Day 757 (n=1) | 20.3 (NA) — NA - Not available, standard deviation is not evaluable when n=1
  Day 1177 (n=1): number analyzed (Participants) | 1
  Day 1177 (n=1) | 31.4 (NA) — NA - Not available, standard deviation is not evaluable when n=1

4. Secondary Outcome: Changes From Baseline in Physical Function Reported by Patients
Description: Self-reported physical function was assessed by a newly developed patient reported outcome named sporadic inclusion body myositis (sIBM) functional assessment (sIFA). The sIFA consists of 11 items scored on an 11 point numerical rating scale from 0 (no difficulty) to 10 (unable to do) across 3 domains: upper body functioning, lower body functioning and general functioning. Participants completed the assessment where the recall period was the past week prior to completing the patient reported outcome (PRO). The total score on the sIFA scale ranges from 0 (minimum) to 110 (maximum). Higher values represent a worse outcome. A positive change from baseline indicates deterioration. Due to the no-signal this analysis was cancelled.
Time Frame: Baseline, Week 104
Population: Due to the early study termination and the small sample size in this open-label trial, this PRO analysis was cancelled.
Arm/Group | BYM338
Number analyzed (Participants) | 0

5. Secondary Outcome: Changes From Baseline in Muscle Strength.
Description: Quadriceps muscle strength was measured, Quadriceps Quantitative Muscle Testing (QMT) by portable fixed dynamometry (PFD). A negative change from baseline indicates deterioration
Time Frame: Baseline, Day 1, 113, 169, 365, 533, 729
Population: Pharmacodynamics (PD) analysis set: Patients with available PD data and no protocol deviations with relevant impact on PD data
Measure: Mean (Standard Deviation); unit: Newtons
Arm/Group | BYM338
Number analyzed (Participants) | 10
Newtons
  Quadriceps score left side Day 1: number analyzed (Participants) | 9
  Quadriceps score left side Day 1 | 0 (0)
  left side Day 113: number analyzed (Participants) | 9
  left side Day 113 | -5.80 (28.160)
  left side Day 169: number analyzed (Participants) | 8
  left side Day 169 | -5.95 (26.587)
  left side Day 365: number analyzed (Participants) | 9
  left side Day 365 | -9.51 (28.149)
  left side Day 533: number analyzed (Participants) | 7
  left side Day 533 | -25.77 (21.321)
  left side Day 729: number analyzed (Participants) | 1
  left side Day 729 | 178.26 (NA) — NA- Not available, standard deviation is not evaluable when n=1
  Quadriceps score Right side Day 1: number analyzed (Participants) | 9
  Quadriceps score Right side Day 1 | 0 (0)
  Right side Day 113 | -4.83 (29.904)
  Right side Day 169: number analyzed (Participants) | 9
  Right side Day 169 | -22.81 (18.784)
  Right side Day 365: number analyzed (Participants) | 9
  Right side Day 365 | -11.63 (47.141)
  Right side Day 533: number analyzed (Participants) | 7
  Right side Day 533 | -31.00 (29.173)
  Right side Day 729: number analyzed (Participants) | 1
  Right side Day 729 | -57.66 (NA) — NA - Not available, standard deviation is not evaluable when n=1

6. Secondary Outcome: Changes From Baseline in Muscle Function (Hand-grip and Pinch-grip Dynamometry)
Description: The effect of BYM338 on additional muscle function measures (hand-grip and pinch-grip dynamometry).
Time Frame: Baseline,Day 1, 113, 169, 365, 533, 729
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Newtons
Arm/Group | BYM338
Number analyzed (Participants) | 10
Newtons
  Left hand-grip day 1 | 0 (0)
  Left hand-grip day 113 | 25.58 (37.544)
  Left hand-grip day 169 | 21.36 (43.815)
  Left hand-grip day 365 | -1.42 (47.973)
  Left hand-grip day 533: number analyzed (Participants) | 7
  Left hand-grip day 533 | 2.78 (16.934)
  Left hand-grip day 729: number analyzed (Participants) | 2
  Left hand-grip day 729 | 8.95 (24.034)
  Right hand-grip day 1 | 0 (0)
  Right hand-grip day 113 | 99.59 (184.472)
  Right hand-grip day 169 | 109.05 (214.248)
  Right hand-grip day 365 | 77.46 (160.133)
  Right hand-grip day 533: number analyzed (Participants) | 8
  Right hand-grip day 533 | 53.99 (127.776)
  Right hand-grip day 729: number analyzed (Participants) | 2
  Right hand-grip day 729 | 163.66 (237.402)
  Left hand pinch grip day 1: number analyzed (Participants) | 1
  Left hand pinch grip day 1 | 0 (0)
  Left hand pinch grip day 113 | 7.82 (27.292)
  Left hand pinch grip day 169 | -4.74 (20.210)
  Left hand pinch grip day 365 | -7.30 (35.224)
  Left hand pinch grip day 533: number analyzed (Participants) | 8
  Left hand pinch grip day 533 | -11.40 (21.204)
  Left hand pinch grip day 729: number analyzed (Participants) | 2
  Left hand pinch grip day 729 | -8.41 (46.672)
  Right hand pinch grip day 1 | 0 (0)
  Right hand pinch grip day 113 | -7.55 (26.792)
  Right hand pinch grip day 169 | -9.35 (30.942)
  Right hand pinch grip day 365 | 0.59 (32.094)
  Right hand pinch grip day 533: number analyzed (Participants) | 8
  Right hand pinch grip day 533 | -8.65 (21.491)
  Right hand pinch grip day 729: number analyzed (Participants) | 2
  Right hand pinch grip day 729 | -35.40 (44.820)

7. Secondary Outcome: Changes From Baseline in Muscle Function 6 Minute Walking Distance
Description: The effect of BYM338 on additional muscle function measures (6 minute walking distance). The 6MWD test measured the distance (in meters) that a participant walked in a 6 minute timeframe. A positive change from baseline indicates improvement.
Time Frame: Baseline,Day 1, 113, 169, 365, 533, 729
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | BYM338
Number analyzed (Participants) | 10
Meters
  Day 1 | 0 (0)
  Day 113: number analyzed (Participants) | 9
  Day 113 | -1.56 (13.685)
  Day 169: number analyzed (Participants) | 9
  Day 169 | -7.41 (12.463)
  Day 365: number analyzed (Participants) | 7
  Day 365 | -8.97 (15.763)
  Day 533: number analyzed (Participants) | 6
  Day 533 | -16.99 (22.382)
  Day 729: number analyzed (Participants) | 1
  Day 729 | -17.86 (NA) — NA - Not available, standard deviation is not evaluable when n=1

8. Secondary Outcome: Change From Baseline of Thigh Muscle Volume (TMV) by MRI Scan
Description: Thigh Muscle Volume (TMV) change was evaluated by a responder analysis. Patients whose loss of muscle TMV by MRI was equal or more than 2% at Week 8 and 16 were considered responders
Time Frame: Baseline, Day 1, 57, 113
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Percentage Change
Arm/Group | BYM338
Number analyzed (Participants) | 10
Percentage Change
  Day 1 | 0 (0)
  Day 57 | 4.14 (4.250)
  Day 113 | 4.51 (6.300)

9. Secondary Outcome: Pharmacokinetics (PK) Parameter of Cmax
Description: To obtain pharmacokinetic data from multiple i.v. dosing of BYM338 in this patient population. Pre-dose, 30 mins & 4 hours post-dose on Day 1.
Time Frame: Day 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | BYM338
Number analyzed (Participants) | 9
ug/mL | 278 (62.6)

10. Secondary Outcome: Time to Reach the Maximum Concentration After Drug Administration (Tmax)
Description: The time to reach the maximum concentration after drug administration
Time Frame: Day 1
Population: as for outcome 3
Measure: Median (Full Range); unit: hr
Arm/Group | BYM338
Number analyzed (Participants) | 9
hr | 0.744 (NA) [0.648 to 4.73]

ADVERSE EVENTS:
Time Frame: period up to 104 weeks
Groups:
- BYM338 10mg/kg i.v.: BYM338 10mg/kg i.v.
Arm/Group | BYM338 10mg/kg i.v.
Serious Adverse Events (participants affected / at risk) | 2/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BYM338 10mg/kg i.v. (N=10)
Anaemia (Blood and lymphatic system disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Tachyarrhythmia (Cardiac disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Iron deficiency (Metabolism and nutrition disorders) | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BYM338 10mg/kg i.v. (N=10)
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 6
Frequent bowel movements (Gastrointestinal disorders) | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 1
Oedema peripheral (General disorders) | 3
Peripheral swelling (General disorders) | 1
Cellulitis (Infections and infestations) | 1
Fungal skin infection (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 3
Avulsion fracture (Injury, poisoning and procedural complications) | 1
Bone contusion (Injury, poisoning and procedural complications) | 1
Concussion (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Corneal abrasion (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 9
Laceration (Injury, poisoning and procedural complications) | 1
Ligament sprain (Injury, poisoning and procedural complications) | 3
Limb injury (Injury, poisoning and procedural complications) | 1
Scratch (Injury, poisoning and procedural complications) | 1
Skin abrasion (Injury, poisoning and procedural complications) | 5
Tibia fracture (Injury, poisoning and procedural complications) | 1
Mammogram abnormal (Investigations) | 1
Natural killer cell count increased (Investigations) | 1
Vitamin D decreased (Investigations) | 1
Weight decreased (Investigations) | 1
Abnormal loss of weight (Metabolism and nutrition disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 2
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1
Gout (Metabolism and nutrition disorders) | 2
Iron deficiency (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 9
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dementia (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 2
Hypogeusia (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Breast hyperplasia (Reproductive system and breast disorders) | 1
Cervical polyp (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Acne (Skin and subcutaneous tissue disorders) | 5
Blister (Skin and subcutaneous tissue disorders) | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1
Papule (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 3
Skin hypertrophy (Skin and subcutaneous tissue disorders) | 1
Thrombophlebitis superficial (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.